CLINICAL TRIAL: NCT02191605
Title: Computer-based Screening, Brief Intervention, and Referral to Treatment (SBIRT) for Marijuana Use in Pregnancy: Planning a Stage II Trial
Brief Title: Computer-delivered Screening & Brief Intervention for Marijuana Use in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34DA036788 (NIH); 1R34DA036788 (NIH)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Marijuana Use; Pregnancy
Keywords: Computerized Brief Intervention
MeSH Terms: conditions — Marijuana Use

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- electronic SBIRT (eSBIRT) (Experimental): Participants in this condition will receive empathic exploration of their thoughts regarding marijuana use, provision of information on possible consequences of marijuana use during pregnancy and potential benefits of changing use (with permission), normed feedback, use of Motivational Interviewing techniques to elicit their own reasons for change, video testimonials modeling successful change, and information on change methods with optional goal setting.
  Interventions: Behavioral: eSBIRT
- Tailored texting (Experimental): Participants in this condition will chose the frequency and time of text messages that will continue until childbirth or the participant opts out. The text messages will be a mix of marijuana targeted content (without directly referring to marijuana in a way that implies use by the participant) and general content related to healthy pregnancy; using appropriate humor and tips for community resources. Tailoring will focus on gestational age, self-efficacy, and social support.
  Interventions: Behavioral: Tailored texting
- eSBIRT & texting (Experimental): Participants in this arm will receive both the computerized intervention and tailored text messaging intervention as described in the eSBIRT and Tailored texting arms.
  Interventions: Behavioral: eSBIRT; Behavioral: Tailored texting
- Assessment only (No Intervention): Participants in the arm will participant in screening and the baseline assessment conducted on the computer only. They will not receive an intervention.
- Screening only (No Intervention): Participants in this arm of the study will only answer the screening questions and will not be asked the baseline assessment or participate in an intervention.

INTERVENTIONS:
Behavioral: eSBIRT — A single 20 minute interactive computer-delivered intervention designed to promote motivation to change prenatal marijuana use, without presuming the participant to be currently using marijuana while pregnant.
  Arms: eSBIRT & texting; electronic SBIRT (eSBIRT)
Behavioral: Tailored texting — Group text messaging software from Trumpia, Inc. will be used to create the tailored text messages that will be sent to participants assigned to this intervention. Text messages will sent after the initial study participation visit until childbirth or participant opts out of receiving them.
  Arms: Tailored texting; eSBIRT & texting

SUMMARY:
Marijuana is by far the mostly commonly used illicit drug during pregnancy, and prenatal exposure to marijuana can have lasting negative effects. However, current answers to this problem are failing to reach most women who use marijuana while pregnant. This project will develop and begin testing two technology-based, highly practical interventions that could reduce the number of children who are prenatally exposed to marijuana.

DETAILED DESCRIPTION:
There are at present no evidence-based interventions for marijuana use during pregnancy, despite its being by far the most commonly used illicit drug during pregnancy (particularly among African-American women), and despite growing evidence that it may have a range of long-term cognitive and neurobehavioral consequences. This R34 clinical trial planning grant therefore proposes the development and preliminary validation of two high- reach and mutually compatible technology-based interventions for marijuana use during pregnancy. The first, a theory-based, synchronous, and highly interactive computer-delivered brief intervention, will be based on an emerging knowledge base regarding key elements of efficacious technology-delivered interventions. The second intervention, a series of tailored text messages, will build on the rich literature regarding key tailoring elements. These interventions will be developed and refined with input from pregnant women who report active use of marijuana, as well as from health care providers. They will subsequently be tested-alone and in combination-in a pilot randomized trial involving 80 women actively using marijuana during pregnancy. This Stage I pilot work would set the stage for a confirmatory Stage II trial. It would also produce the first high-reach brief interventions for marijuana use during pregnancy. If effective, these approaches could have a substantial population impact on marijuana use among pregnant women, with potential for lifelong improved outcomes for both mother and child.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age
* 20 weeks or less gestation
* intention to carry pregnancy to term
* self-reported marijuana use in month before pregnancy
* own a cell phone and willingness to receive text messages
* gives consent to access medical records for collection of birth outcome data

Exclusion Criteria:

* frank cognitive impairment or psychosis
* not able to communicate in English
* not planning to deliver at a Detroit Medical Center (DMC) hospital
* previous or current participant in a study conducted by Dr. Ondersma
* Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Perinatal Research Branch participant.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electronic SBIRT (eSBIRT) | Tailored Texting | eSBIRT & Texting | Assessment Only | Screening Only
Started | 15 | 15 | 15 | 8 | 7
Completed Intervention Portion | 15 | 15 | 15 | 8 | 7
Completed (Completed postpartum follow-up) | 6 | 11 | 8 | 5 | 3
Not Completed | 9 | 4 | 7 | 3 | 4
Not completed — Lost to Follow-up | 9 | 4 | 7 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electronic SBIRT (eSBIRT) | Tailored Texting | eSBIRT & Texting | Assessment Only | Screening Only | Total
Number analyzed (Participants) | 15 | 15 | 15 | 8 | 7 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (5.9) | 23.5 (3.7) | 27.2 (5.4) | 22.6 (3.2) | NA (NA) — Only verified 18 and older during screening. Continuous measure of age asked during assessment. | 24.6 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 8 | 7 | 60
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 15 | 8 | 7 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 12 | 15 | 8 | 5 | 51
  White | 1 | 2 | 0 | 0 | 1 | 4
  More than one race | 3 | 1 | 0 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
ASSIST marijuana score [Median (Inter-Quartile Range); unit: scores on a scale] — The Alcohol Smoking and Substance Involvement Screening Test (ASSIST) was developed by the World Health Organization (WHO) and is used to detect and manage substance use and related problems. For this measure the sum of all the marijuana related items was calculated for each participant. We reported the median score for each intervention arm group. Scores on the marijuana subscale range from 0 to 33. Scores of 0 to 3 present low risk; 4 - 26 moderate risk (at risk of health & other problems from current pattern of use); and 27 - 33 high risk (severe problems & likely to be dependent).
  scores on a scale | 9 [0 to 12] | 9 [4 to 16] | 6 [5 to 12] | 6 [0.5 to 11] | NA [NA to NA] — ASSIST not given during screening | 8 [2 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Abstinent From Marijuana for the 7 Days Prior to Delivery
Description: Marijuana use will be measured at the time of delivery of their infant by self-report (TimeLine Follow Back interview - TLFB) and urine analysis. This will represent the number of participants who abstinent (reported no marijuana use and had a negative toxicology urine screen) from marijuana for the 7 days prior to delivery.
Time Frame: self-reported use during 7 days prior to delivery of their baby
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic SBIRT (eSBIRT) | Tailored Texting | eSBIRT & Texting | Assessment Only | Screening Only
Number analyzed (Participants) | 6 | 7 | 7 | 3 | 3
Participants | 6 | 7 | 6 | 3 | 2

2. Primary Outcome: Number of Participants Abstinent From Marijuana for the 90 Days Prior to Delivery
Description: Marijuana use will be measured at the time of delivery of their infant by self-report (TimeLine Follow Back interview - TLFB) and hair toxicology analysis. This will represent the number of participants who were abstinent (reported no marijuana use and had a negative hair toxicology results) from marijuana for the 90 days prior to delivery.
Time Frame: self-reported use during 90 days prior to delivery of their baby
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic SBIRT (eSBIRT) | Tailored Texting | eSBIRT & Texting | Assessment Only | Screening Only
Number analyzed (Participants) | 3 | 6 | 2 | 2 | 3
Participants | 2 | 5 | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: remainder of the pregnancy (24-20 weeks)
Arm/Group | Electronic SBIRT (eSBIRT) | Tailored Texting | eSBIRT & Texting | Assessment Only | Screening Only
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT02191605/Prot_SAP_000.pdf